CLINICAL TRIAL: NCT06390527
Title: Optimization of Ultrasound Sheer Wave Elastography for the Evaluation of Peripheral Nerve Disorders
Brief Title: Ultrasonography in Diagnosis of Polyneuropathy
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: USpolyneuropathy
Record Dates: First submitted 2024-01-03; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Polyneuropathies
MeSH Terms: conditions — Polyneuropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main goal of this trial is to establish recommendations for clinical practice that enhance the reliability, accessibility and convenience of sheer wave elastography as a routine diagnostic test for diverse peripheral neuropathies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Clinical signs of particular polyneuropathy not explained by other causes

Exclusion Criteria:

* Entrapment or compression neuropathies
* Nerve trauma
* The diagnosis of vasculitic neuropathy, neuralgic amyotrophy, diabetic radiculo-plexo-neuropathy, hereditary neuropathy with liability to pressure palsies and motor neuron disorders including monomelic amyotrophy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral polyneuropathy recruited from the electronic database at the institute of Clinical Neurophysiologym Division of Neurology, University Medical Centre Ljubljana, Slovenia, and distributed in groups with different types of polyneuropathy.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Clinical examination | Through study completion, an average 2 years.
  1) Myotatic reflexes (biceps, triceps, finger flexors, patellar, Achilles, deep abdominal): 1-absent, 2-reduced or 3-present with facilitation.
  1. Muscle atrophy: 1-no atrophy, 2-mild, 3-moderate or4-severe atrophy
  2. Muscle strength of lower and upper limbs with Medical Research Council (MRC) scale (0-5/5): shoulder abduction, elbow flexion and extension, wrist flexion and extension, fingers flexion, extension and abduction, hip flexion, extension, abduction and adduction, knee flexion and extension, ankle dorsal flexion, plantar flexion, eversion and inversion, thumb flexion and extension.
  3. Touch sensation in all dermatomes with cotton wool: 1-normal sensation, 2-mild, 3-severe or 4-absent.
Electrodiagnostic studies | Through study completion, an average 2 years.
  1. Motor nerve conduction studies in median, ulnar, radial, fibular and tibial: distal motor latency, compound muscle action potential (CMAP) amplitude, duration and area, conduction velocity.
  2. Sensory nerve conduction studies in median, ulnar, superficial radial, superficial fibular and sural nerve: latency, sensory nerve action potential (SNAP) amplitude and velocity
Ultrasonography | Through study completion, an average 2 years.
  Cross-sectional area (CSA) and shear-wave velocity (SV) of:
  1. median nerve at wrist, forearm, elbow and upper arm
  2. ulnar nerve at wrist, forearm, elbow and upper arm
  3. radial nerve at elbow and upper arm
  4. vagus nerve
  5. brachial plexus (C5,6 and 7)
  6. fibular nerve at capitulum fibulae and popliteal fossa
  7. tibial nerve at the medial malleolus and popliteal fossa
  8. sciatic nerve
  9. sural nerve
Patient history | Through study completion, an average 2 years.
  1. demographic data: sex, date of birth, height, weight
  2. symptoms duration (months), symptoms, therapy